CLINICAL TRIAL: NCT00046059
Title: Genetic Analysis of Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000058; 00-HG-0058
Record Dates: First submitted 2002-09-18; First posted 2002-09-19 (Estimated); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: ADHD
Keywords: Linkage; Gene Identification; Hyperactivity; Natural History; Attention Deficit Hyperactivity Disorder; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADHD: Children aged 7-17 with ADHD and their families.

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is the most common behavioral disorder in childhood, affecting 3-5% of children between the ages of 7 and 17. Family studies suggest that there is a genetic component to ADHD. Scientists believe that it is a complex disorder in which two or more genes may be involved.

Potentially eligible families will be asked to give written consent to participate and will be asked to complete questionnaires for each member in the family. In addition, an interview will be administered to the parent of minors enrolled in the study to determine their eligibility for being in the study. This screening tool is computerized and will take approximately 45 minutes to administer per child.

Once screenings are completed, a blood collection kit will be sent to the family to take to their local medical care provider, have blood samples drawn and sent to NIH. There is no cost to the family to participate. We would like to enroll entire families, with both parents and all children.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) is one of the most common childhood

disorders and the most common childhood neurodevelopmental behavioral disorder. Symptoms include difficulty staying focused (inattention), difficulty controlling behavior (impulsivity), and hyperactivity. Symptoms typically develop between six and 12 years of age, and frequently persist into adulthood, with serious life-long health and social consequences. Affected children are at increased risk for poor educational achievement, low income, underemployment, legal difficulties, and impaired social relationships. The general belief is that ADHD is caused by a combination of genetic and environmental factors.

The main objective of the study is to conduct genetic and behavioral studies that will closely

characterize the genetic influences in diagnosis, prognosis, severity, and pharmacological

response in ADHD patients. Since the start of the study in 2000, research has contributed to the understanding of the innate susceptibility of ADHD and associated comorbidities; the interaction of genetic, demographic, and environmental factors underpinning the risk of developing ADHD; the extent to which these factors shape the response of ADHD patients to pharmacological interventions (pharmacogenetics); the over-representation of functional and ontological genebased networks implicated in determining synapse structure; and the use of advanced geneticepidemiological models with potential for use in clinical practice (translational genomics). The most significant research finding occurred in 2010, when the study team identified LPHN3, a key gene involved in the etiology of ADHD and comorbid conditions in one of the previously identified regions of strong genetic signal in chromosome 4q13.2.

In order to provide power for the study s statistical analyses, the upper enrollment goal is 4,000 participants. Although the study has several small and genetically distinct cohorts, the majority of subjects come from the United States of America population through outreach recruitment efforts. Recruitment has been very successful and the large cohort numbers provide support for identification of genetic components related to the diagnosis of ADHD. Recent efforts have focused on identifying new areas of the genome associated with ADHD, and identifying genetic (coding and non-coding) variations implicated in the etiology and clinical manifestations of ADHD. A primary aim of the study is to correlate genetic and biological markers for diagnosis and prognosis of ADHD identified through the use of state of the art genomics, which includes enome-wide association studies, linkage analysis, whole genome and exome sequencing, and targeted gene capture in cosmopolitan and isolated populations. As the current diagnosis of ADHD is based on subjective observations, one of the main goals of the study is to develop a more definitive system to diagnose ADHD and to assess and predict prognosis.

ELIGIBILITY:
* INCLUSION CRITERIA:

This study will enroll families with the following characteristics:

1. Families with children, seven through 17 years of age, diagnosed with ADHD (defined as the proband for the study).
2. The probands siblings, either affected with ADHD (concordant) or unaffected (discordant), seven years of age and above, including adult siblings.
3. The parents, both mothers and fathers, of enrolled probands.
4. The study will enroll both male and female probands of any ethnic background and race. The prevalence of ADHD is higher in males than in females, so we would expect to have a higher number of male probands than female probands. Both male and female siblings and male and female parents of probands will be enrolled.
5. Adults who are or may be unable to provide informed consent will be excluded.
6. Probands with one parent affected with ADHD or with neither parent affected with ADHD are eligible. Probands from bilineal families, families with both parents affected with ADHD, will be excluded for statistical reasons.

Additional inclusion criteria for the study include:

1. Ability to read and understand spoken English, since the questionnaires, scales, and interviews that we have license to use in this study are in English.

EXCLUSION CRITERIA:

Some conditions can confound the diagnosis of ADHD. Probands with the following conditions will be excluded from enrollment or will be withdrawn from the study if the condition is discovered subsequent to enrollment:

* Prematurity
* Neurological conditions
* Cardiac surgery
* Prenatal drug exposure
* Hydrocephaly
* Mental Retardation (IQ<80)
* Known genetic syndromes
* Known CNS disorders
* Known lead toxicity
* Tourette Disorder
* Obsessive-Compulsive Disorder
* Major Depression on both proband and affected sibling
* Pervasive Developmental Disorder
* Age under 7 years old
* Autism
* Other Psychoses
* Post Traumatic Stress Disorder
* Language Disorder (if known)
* Severe Sensory Impairment (visual and hearing)

Probands with the following conditions may be included, but the conditions will be noted during statistical analysis:

* Oppositional Defiant Disorder
* Conduct Disorder
* Tic Disorder
* Obsessive/Compulsive Symptoms
* Anxiety/Phobias
* Learning Disabilities

Ages: 7 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Families with children, seven through 17 years of age, diagnosed with ADHD (defined as the proband for the study). 2. The probands siblings, either affected with ADHD (concordant) or unaffected (discordant), seven years of age and above, including adult siblings. 3. The parents, both mothers and fathers, of enrolled probands.
Sampling Method: Non-Probability Sample
Enrollment: 3481 (Actual)
Dates: Start 2000-02-08 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
ADHD | Ongoing
  The main objective of the study is to conduct genetic and behavioral studies that will closely characterize the genetic influences in diagnosis, prognosis, severity, and pharmacological response in ADHD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Acosta, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - University of California, Irvine Medical Center, Orange, California
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided
pending

REFERENCES:
- [Background] Anderson JC, Williams S, McGee R, Silva PA. DSM-III disorders in preadolescent children. Prevalence in a large sample from the general population. Arch Gen Psychiatry. 1987 Jan;44(1):69-76. doi: 10.1001/archpsyc.1987.01800130081010. PMID 2432848
- [Background] Biederman J, Faraone S, Milberger S, Guite J, Mick E, Chen L, Mennin D, Marrs A, Ouellette C, Moore P, Spencer T, Norman D, Wilens T, Kraus I, Perrin J. A prospective 4-year follow-up study of attention-deficit hyperactivity and related disorders. Arch Gen Psychiatry. 1996 May;53(5):437-46. doi: 10.1001/archpsyc.1996.01830050073012. PMID 8624187
- [Background] Faraone SV, Biederman J, Chen WJ, Milberger S, Warburton R, Tsuang MT. Genetic heterogeneity in attention-deficit hyperactivity disorder (ADHD): gender, psychiatric comorbidity, and maternal ADHD. J Abnorm Psychol. 1995 May;104(2):334-345. doi: 10.1037/0021-843X.104.2.334. PMID 7790635
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-HG-0058.html